CLINICAL TRIAL: NCT05936684
Title: Breathing and Decision-Making: an FMRI Study Investigating the Link Between Slow Breathing and Risky Decision-Making
Brief Title: Breathing and Decision-Making
Acronym: ProlEx-MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Charite University, Berlin, Germany (Other); German Center for Diabetes Research (Other); Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Prof. Dr., German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ProlEx-MRI
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Quality of Life; Behavior; Stress, Psychological
Keywords: Breathing; Relaxation; Decision-Making; Stress Management
MeSH Terms: conditions — Behavior; Stress, Psychological; Respiratory Aspiration | interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of ProlEx breathing on decision-making if applied before the Eupnea condition (Experimental): Intervention (behavioral): Block 1: ProlEx, Block 2: Eupnea/Control during decision-making
  Interventions: Behavioral: Breathing with prolonged exhalation (ProlEx) during risky decision-making; Behavioral: Normal breathing (Eupnea/Control) during risky decision-making
- Effect of Eupnea breathing on decision-making if applied before the ProlEx condition (Experimental): Intervention (behavioral): Block 1: Eupnea/Control, Block 2: ProlEx during decision-making
  Interventions: Behavioral: Breathing with prolonged exhalation (ProlEx) during risky decision-making; Behavioral: Normal breathing (Eupnea/Control) during risky decision-making

INTERVENTIONS:
Behavioral: Breathing with prolonged exhalation (ProlEx) during risky decision-making — 20 min divided in 3 blocks of slow, 0.1 Hz breathing (6 cycles per minute) with an inhalation-to-exhalation ratio of 2:8. Cue-assisted breathing (same across participants) and performance of a risky decision-making task (Tom et al., 2007) in the magnetic resonance imaging (MRI) scanner with simultaneous acquisition of physiological and pupil data.
  Other Names: ProlEx (decision-making); Slow Breathing
Behavioral: Normal breathing (Eupnea/Control) during risky decision-making — 20 min divided in 3 blocks of normal breathing (expected range: 0.16-0.33 Hz, i.e., 10-20 per min), Cue-assisted breathing (individually adapted) and performance of a risky decision-making task (Tom et al., 2007) in the MRI scanner with simultaneous acquisition of physiological and pupil data.
  Other Names: Eupnea (decision-making); Normal Breathing

SUMMARY:
The study aims to investigate how slow breathing with prolonged exhalation (i.e., ProlEx breathing) modulates decision-making under risk in healthy participants. To do this, a short-term breathing intervention is combined with a decision-making paradigm while neural, physiological, and behavioral data are recorded.

DETAILED DESCRIPTION:
This interventional study investigates the modulatory effect of slow breathing with prolonged exhalation (i.e., ProlEx breathing) on decision-making under risk. Using functional magnetic resonance imaging (fMRI), the researchers seek to identify brain regions influenced by the breathing intervention during the decision-making task.

Sixty healthy participants will be invited to perform ProlEx breathing during a risky decision-making task. After initial preparations, each individual's spontaneous breathing rhythm will be determined (i.e., Eupnea, control condition). This step is to i) ensure a natural breathing pace for each participant and ii) incorporate cue-assisted breathing into the control condition to allow comparability across conditions. To further investigate the effect of ProlEx on sympathovagal tone, physiological measures of respiration, electrocardiogram, pulse, electrodermal activity, and pupil are acquired. During scanning, the participant will perform a decision-making task based on the paradigm by Tom et al. (2007). The breathing intervention is applied simultaneously with continuous cue-assisted breathing for both conditions (Eupnea, ProlEx) throughout the duration of the task. The experiment follows a block design with counterbalanced orders to control for confounding effects. After completion of the scans, the participants fill out additional questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Normal vision (no glasses or contact lenses required)

Exclusion Criteria:

* Smokers
* Extreme athletes
* Extensive lung function (e.g., professional musician, abnoedivers)
* Excessive stress
* Former or current physical or psychological illness (e.g., lung diseases)
* Current or previous medication within 2 weeks before the appointment
* Left-handedness
* Claustrophobia
* Tinnitus
* Non-removable metal parts or implants inside or on the body (e.g., hip replacements, copper IUD)
* Non-removable ferromagnetic objects inside or on the body (e.g., joint replacements)
* Non-removable magnetic objects inside or on the body (e.g., artificial eye)
* Large tattoos
* Young (>18 years) or old (>40 years) subjects
* Over- or underweight (BMI <18 or >25 kg/m2)
* Pregnancy
* Abnormal circadian rhythm (e.g., during shift work)
* Excessive alcohol consumption
* Illegal drug consumption within 2 weeks before the appointment
* Missing consent to participate
* Missing consent to receive incidental findings (MRI)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Behavior: Risk propensity | 1 year
  Risk propensity, i.e., the willingness to accept or reject a risky mixed gamble in an adapted paradigm based on Tom et al. (2007); assessed using response options "strongly accept", "weakly accept", "weakly reject", "strongly reject"
Brain: blood-oxygen-level-dependent (BOLD) signal changes | 1 year
  BOLD signal changes on a whole-brain level and in predefined regions of interest assessed using fMRI
Body: Heart-rate variability | 1 year
  Low-frequency and high-frequency heart rate variability (LF-HRV and HF-HRV, respectively); assessed using an electrocardiogram (ECG) and pulse oximetry
Body: Pupil | 1 year
  Miosis/mydriasis, i.e., changes in pupil dilation; assessed with eye tracking
Body: Electrodermal activity | 1 year
  Tonic electrodermal activity (EDA); assessed using a galvanic skin response module

SECONDARY OUTCOMES:
Questionnaire assessing depression: "Beck Depression Inventory" (BDI) | 1 year
  The depression scale (self-report) will be assessed using Beck Depression Inventory (BDI) (Hautzinger et al., 1994). The questionnaire consists of 21 questions, with each item corresponding to a value ranging from 0 to 3. Higher total scores indicate more severe depressive symptoms. A total score of 0-13 is considered minimal, 14-19 mild, 20-28 moderate, and 29-63 severe.
Questionnaire assessing personality traits: "Big Five Inventory" (BFI-10) | 1 year
  Personality traits (self-report) will be assessed using the Big Five Inventory (BFI-10) (Rammstedt et al., 2013). The BFI-10 is a 10-item scale measuring the Big Five personality traits Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness. Ten items are answered on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree".
  Scoring of the BFI-10 scales (R = item is reverse-scored): Extraversion: 1R, 5; Agreeableness: 2, 7R; Conscientiousness: 3R, 8; Neuroticism: 4R, 9; Openness to Experience: 5R, 10.
  Individuals who score high on the BFI-10 tend to exhibit certain qualities associated with each of the personality traits. The score can range from a minimum of 2 to a maximum of 10 points for each of the personality traits.
Questionnaire assessing impulsivity: "Barratt Impulsivity Scale" (BIS-15) | 1 year
  Impulsivity (self-report) will be assessed using the Barratt Impulsivity Scale (BIS-15) (Meule et al., 2011). This scale is a questionnaire consisting of 15 items scored from 1 to 4 with 1 = rarely / never, 2 = sometimes, 3 = often, and 4 = almost always / always. Scores range from 15 to 60, with higher scores reflecting greater impulsiveness.
Questionnaire assessing approach-avoidance behavior: "Behavioral Inhibition System/Behavioral Approach System" (BIS/BAS) | 1 year
  Approach-avoidance behavior (self-report) will be assessed using the Behavioral Inhibition System/Behavioral Approach System (BIS/BAS) (Strobel et al., 2001).
  The BIS/BAS scale is a 24-item self-report questionnaire designed to measure two motivational systems. The behavioral inhibition system (BIS), which corresponds to the motivation to avoid aversive outcomes, has 7 items with a total score ranging from 7 to 28 points. The behavioral activation system (BAS), which corresponds to the motivation to approach goal-oriented outcomes,has 13 items with a total score ranging from 13 to 52 points. Four items act as filler items. Participants respond to each item using a 4-point Likert scale: 1 (very true for me), 2 (somewhat true for me), 3 (somewhat false for me), and 4 (very false for me). Total scores are calculated for BIS and BAS, with a higher score corresponding to higher behavioral inhibition and activation, respectively.
Questionnaire assessing self-control: "Brief Self-Control Scale" (BSCS) | 1 year
  Self-control (self-report) will be assessed using the Brief Self-Control Scale (BSCS) (Sproesser et al., 2011). The BSCS measures trait self-control via items with a 5-point Likert scale, where 1 refers to 'not at all' and 5 to 'extremely'. Scores range from 13 to 65. Higher scores represent higher levels of self-control.
Questionnaire assessing interoceptive awareness: "Multidimensional Assessment of Interoceptive Awareness" (MAIA-2) | 1 year
  Interoceptive Awareness (self-report) will be assessed using the "Multidimensional Assessment of Interoceptive Awareness" (MAIA-2) (Mehling et al., 2018). The MAIA assesses multidimensional aspects of self-reported interoception and includes 37 items using a six-point Likert scale (0 never, 5 always). Higher scores equate to higher awareness of bodily sensation.
  The results from the MAIA-2 focus on the individual scale scores (Mehling et al., 2012).
Questionnaire assessing affect: "Positive and Negative Affect Scale" (PANAS) | 1 year
  Affect (self-report) will be assessed using the Positive and Negative Affect Scale (PANAS) (Janke et al., 2014). The PANAS is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Score: the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: Add the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 10 to 50, with lower scores representing lower levels of negative affect.
Questionnaire assessing stress: "Perceived Stress Questionnaire" (PSQ) | 1 year
  Stress (self-report) will be assessed using the Perceived Stress Questionnaire (PSQ) (Fliege et al., 2001). The PSQ a self-report questionnaire that consists of 20 items. Each item is rated on a 4-point Likert scale of 1 to 4. Total scores range from 20 to 80. Higher scores indicate greater levels of stress.
Questionnaire assessing self-efficacy: "General Self-Efficacy Scale" (GSE) | 1 year
  Self-efficacy (self-report) will be assessed using the General Self-Efficacy Scale (GSE) (Schwarzer et al., 1997). The GSE is a 10-item scale with a score for each item ranging from 1 to 4. Total scores range from 10 to 40. Higher scores indicate higher self-reported self-efficacy.
Questionnaire assessing anxiety: "State-Trait Anxiety Inventory" (STAI-T) | 1 year
  Trait anxiety (self-report) will be assessed using the State-Trait Anxiety Inventory (STAI-T) (Grimm et al., 2009). The State-Trait Anxiety Inventory (STAI-T) is a 20-item scale with a score for each question ranging from 0 to 3. Total scores range from 0 to 60. Higher scores indicate higher levels of anxiety.
Questionnaire assessing mentall well-being: "Warwick-Edinburgh Mental Well-Being Scale" (SWEMWBS) | 1 year
  Mental well-being (self-report) will be assessed using the Warwick-Edinburgh Mental Well-Being Scale, short version (SWEMWBS) (Lang et al., 2017). The WEMWBS is scored by summing the responses to each of the 14 items on a 1 to 5 Likert scale. Total scores can range from a minimum of 14 to a maximum of 70 points. Higher scores are associated with higher levels of mental well-being.
Body: Eye gaze | 1 year
  Eye fixation points analysed using eye-tracking data

CONTACTS AND LOCATIONS:
Overall Officials: Soyoung Q Park, Prof. Dr., Principal Investigator — German Institute of Human Nutrition
Locations (1):
- German Institute of Human Nutrition, Nuthetal, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fliege, H., Rose, M., Arck, P., Levenstein, S. & Klapp, B. F. (2001). Validierung des Perceived Stress Questionnaire (PSQ) an einer deutschen Stichprobe. Diagnostica, 47, 142-152.
- [Background] Grimm, J. State-trait-anxiety inventory nach Spielberger. Deutsche Lang- und Kurzversion. Methodenforum der Universität Wien: MF-Working Paper (2009).
- [Background] Hautzinger M. [The Beck Depression Inventory in clinical practice]. Nervenarzt. 1991 Nov;62(11):689-96. German. PMID 1770969
- [Background] Janke, S., & Glöckner-Rist, A. (2014). "Deutsche Version der Positive and Negative Affect Schedule (PANAS)" in Zusammenstellung sozialwissenschaftlicher Items und Skalen, GESIS (Mannheim, Germany). doi.org/10.6102/zis146
- [Background] Lang, G. & Bachinger, A. Validation of the German Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) in a community-based sample of adults in Austria: a bi-factor modelling approach. J Public Health 25, 135-146 (2017)
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Meule, A., Vögele, C. & Kübler, A. Psychometrische Evaluation der deutschen Barratt Impulsiveness Scale - Kurzversion (BIS-15). Diagnostica 57, 126-133 (2011).
- [Background] Rammstedt, B., Kemper, C.J., Klein, M.C., Beierlein, C., & Kovaleva, A. (2013). Eine kurze Skala zur Mes-sung der fünf Dimensionen der Persönlichkeit. Methoden, Daten, Analysen, 7(2), S. 233-249
- [Background] Schwarzer, R., Bäßler, J., Kwiatek, P., Schröder, K., & Zhang, J. X. (1997). The assessment of optimistic self-beliefs: comparison of the German, Spanish, and Chinese versions of the general self-efficacy scale. Applied Psychology, 46(1), 69-88.
- [Background] Tom SM, Fox CR, Trepel C, Poldrack RA. The neural basis of loss aversion in decision-making under risk. Science. 2007 Jan 26;315(5811):515-8. doi: 10.1126/science.1134239. PMID 17255512